CLINICAL TRIAL: NCT05641350
Title: Barlow's unIfied Protocol for emoTional Eating (BITE): a Pre-post Design
Acronym: BITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIBSP-BIT-2022-78
Record Dates: First submitted 2022-11-16; First posted 2022-12-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-03

CONDITIONS: Emotional Eating
MeSH Terms: conditions — Emotional Eating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional eating intervention (Experimental): Emotional eating intervention
  Interventions: Behavioral: Barlow's Unified Protocol
- Waiting list (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Barlow's Unified Protocol — Adaptation of the cognitive-behavioral Barlow's Unified Protocol for emotional eating pattern.
  Arms: Emotional eating intervention

SUMMARY:
This study aims to evaluate the efficacy of a group intervention program, based on the Barlow's protocol, in patients with emotional eating with the aim of improving the emotional eating pattern.

The design is quasi-experimental pre-post with a control group (waiting list) and evaluation of the maintenance of the response after 6 months of the end of the program.

Includes outpatients from the Eating Disorders Unit and the Psychiatry Unit of a Hospital. A sample size of 26 participants is considered in the experimental group, and another 26 more in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients from eating behavior disorder outpatient clinics and psychiatric outpatient clinics.
* Age between 18 and 65 years.
* Score of more than 2.46 on the "emotional eating" subscale of the DEBQ scale

Exclusion Criteria:

* Diagnosis of active Eating Disorder, that is, without at least 6 months of symptomatic remission or that exceed the cut-off point on the EAT-26 scale.
* Patients with severe mental disorder with or without psychotic symptoms (schizophreniform disorders, bipolar spectrum disorders, major depression)
* Patients with some other medical disorder that presents with impulse dysregulation, such as epilepsy, frontal-type dementia...
* Patients with an IQ < 85
* Patients who do not give consent.
* Patients who do not understand or speak Spanish or Catalan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Emotional eating score assessed by the Emotional eating sub-scale of the Dutch Eating Behavior Questionnaire (DEBQ-EE) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided